CLINICAL TRIAL: NCT03198975
Title: Development of a Machine Learning-based Model for Preoperative Prediction of Microvascular Invasion in Hepatocellular Carcinoma
Brief Title: Preoperative Prediction of Microvascular Invasion in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ming Kuang (Other)
Responsible Party: Sponsor-Investigator, Ming Kuang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: HCC10
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: magnetic resonance image features; pathological differentiation; machine learning-based model
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preoperative imaging features: In this project, there is only one study group which comprises of patients with Hepatocellular Carcinoma (HCC) who will undergo preoperative Gd-EOB-DTPA enhanced magnetic resonance image.
  Interventions: Diagnostic Test: Magnetic resonance image

INTERVENTIONS:
Diagnostic Test: Magnetic resonance image — Histologically-diagnosed primary HCC after curative hepatectomy. The magnetic resonance image will be imported into the software ,and the radiomic textural features will be automatically extracted by the Analysis-Kit software.The high-throughput extracted features will be then selected and a prediction model will be developed in the training set in which patients were collected from a retrospective study. In this project, an independent validation set will be collected and used to validate the prediction accuracy of the model.

SUMMARY:
Microvascular invasion (MVI) has been well demonstrated as an unfavorable prognostic factor for hepatocellular carcinoma (HCC), and patients with MVI have a high risk of tumor recurrence after curative hepatectomy. Currently, the diagnosis of MVI is determined on the postoperative histologic examination, which greatly limits its influence on preoperative decision making. Therefore, we constructed this prospective study to develop a machine learning-based model for preoperative prediction of MVI by extracting high-dimensional magnetic resonance (MR) image features.

DETAILED DESCRIPTION:
Histologically-diagnosed primary HCC after curative hepatectomy. The magnetic resonance image will be imported into the imaging management software (GE healthcare Analysis-Kit software),and the tumor lesions will manually delineated by two independent radiologists and then reconstruct into three-dimensional images for feature extraction. The radiomic textural features including grayscale histogram, transform matrix, wavelet transform and filter transformation are automatically extracted by the Analysis-Kit software.The high-throughput extracted features will be then selected by the univariate analysis, and a prediction model will be developed based on machine learning algorithm in a training set in which patients were collected from a retrospective study. And in the present study, an independent validation set will be collected and used to validate the prediction accuracy of the model.

ELIGIBILITY:
Inclusion Criteria:

* Asian patients aged 18～80 years old;
* HCC without macroscopic vascular invasion according to imaging findings;
* Child Pugh A-B stage;
* Receipt of preoperative Gd-EOB-DTPA enhanced MR imaging of the abdomen within one month before surgery;
* Histologically-diagnosed primary HCC after curative hepatectomy;

Exclusion Criteria:

* Combined hepatocellular-cholangiocarcinoma;
* With extra-hepatic metastasis or macrovascular invasion;
* With incomplete clinical and imaging data;
* Non-radical resection;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between June 2017 and July 2017，all patients who will undergo curative resection (R0 resection) at the First Affiliated Hospital of Sun YatSen University in Guangzhou, China, for HCC based on the modified WHO classification of tumors of the digestive system, are considered for inclusion. By the eligibility criteria stated below, MVI presentative rate is 30-42% in chinese HCC population as reported, we retrospectively collected about 80 patients for training and an estimated 40 patients will be needed for validation set of this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
Presence of microvascular invasion | Through patient enrollment completion ,an average of 2 years
  Postoperative histologically confirmed microvascular invasion

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Director — Department of Liver Surgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aerts HJ, Velazquez ER, Leijenaar RT, Parmar C, Grossmann P, Carvalho S, Bussink J, Monshouwer R, Haibe-Kains B, Rietveld D, Hoebers F, Rietbergen MM, Leemans CR, Dekker A, Quackenbush J, Gillies RJ, Lambin P. Decoding tumour phenotype by noninvasive imaging using a quantitative radiomics approach. Nat Commun. 2014 Jun 3;5:4006. doi: 10.1038/ncomms5006. PMID 24892406
- [Result] Zhang YD, Wang Q, Wu CJ, Wang XN, Zhang J, Liu H, Liu XS, Shi HB. The histogram analysis of diffusion-weighted intravoxel incoherent motion (IVIM) imaging for differentiating the gleason grade of prostate cancer. Eur Radiol. 2015 Apr;25(4):994-1004. doi: 10.1007/s00330-014-3511-4. Epub 2014 Nov 28. PMID 25430007
- [Result] Woo S, Lee JM, Yoon JH, Joo I, Han JK, Choi BI. Intravoxel incoherent motion diffusion-weighted MR imaging of hepatocellular carcinoma: correlation with enhancement degree and histologic grade. Radiology. 2014 Mar;270(3):758-67. doi: 10.1148/radiol.13130444. Epub 2013 Oct 30. PMID 24475811
- [Result] Huang YQ, Liang CH, He L, Tian J, Liang CS, Chen X, Ma ZL, Liu ZY. Development and Validation of a Radiomics Nomogram for Preoperative Prediction of Lymph Node Metastasis in Colorectal Cancer. J Clin Oncol. 2016 Jun 20;34(18):2157-64. doi: 10.1200/JCO.2015.65.9128. Epub 2016 May 2. PMID 27138577
- [Result] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733